CLINICAL TRIAL: NCT03004690
Title: Limiting Factors for Wearing Personal Protective Equipment (PPE) in a Health Care Environment Evaluated in a Randomised Study: Source of Errors?
Brief Title: Testing of Personal Protective Equipment (PPE)
Acronym: PPE-Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 23-321
Record Dates: First submitted 2016-12-05; First posted 2016-12-29 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Personal Protective Equipment; Heat Stress
Keywords: biosafety; outbreaks; clinic; personal protective equipment; ergonomics; error rates
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Performance temperature 22°C (Experimental): Participants wearing PPE suit A or PPE suit B perform tests I -IV at 22°C.
  Interventions: Device: PPE Suit A; Device: PPE Suit B
- Performance temperature 28°C (Experimental): Participants wearing PPE suit A or PPE suit B perform tests I -IV at 28°C.
  Interventions: Device: PPE Suit A; Device: PPE Suit B

INTERVENTIONS:
Device: PPE Suit A — In this randomized study following good clinical practice guidelines nineteen study volunteers were recruited to wear one of two different types of randomly allocated PPE suits. Suit A has to be used by randomly selected participants to perform four different tests six times at 22°C on one day and four times at 28°C on another day in the local core facility clinical research center.
  Other Names: Suit A - Tychem F + - 3MTM Mehrwegleichthaube S-655
Device: PPE Suit B — Suit B has to be used by randomly selected participants to perform four different tests six times at 22°C on one day and four times at 28°C on another day in the local core facility clinical research center.
  Other Names: Suit B -- 3MTM JS-Serie Typ 3 Respiratory Protective Suit

SUMMARY:
Pandemics and re-emerging diseases put pressure on the health care system to prepare for patient care and sample logistics requiring enhanced personnel protective equipment (PPE) for health care workers. We generated quantifiable data on ergonomics of PPE applicable in a health care setting by defining error rates and physically limiting factors due to PPE-induced restrictions. Nineteen study volunteers tested randomly allocated head- or full body-ventilated PPE suits equipped with powered-air-purifying-respirators and performed four different tests (two laboratory tutorials, a timed test of selective attention and a test investigating reaction time, mobility, speed and physical exercise) during 6 working hours at 22°C on one day and 4 working hours at 28°C on another day. Error rates and physical parameters (fluid loss, body temperature, heart rate) were determined and ergonomic-related parameters were assessed hourly using questionnaires. Depending on the PPE system the most restrictive factors were: reduced dexterity due to multiple glove layers, impaired visibility by flexible face shields and back pain related to the respirator of the fully ventilated suit. Heat stress and liquid loss were perceived as restrictive at a working temperature of 28°C but not 22°C.

DETAILED DESCRIPTION:
In this randomized study following good clinical practice guidelines nineteen study volunteers were recruited to wear one of two different types of randomly allocated PPE suits (www.randomizer.at) and to perform four different tests six times at 22°C on one day and four times at 28°C on another day in the local core facility clinical research center.

Study participants Recruiting was based on voluntary registration in response to a public announcement. The study was subjected to the local ethical committee review (No. 23-321 ex 10/11) and all persons gave written informed consent according to the Helsinki Declaration. Key lifestyle and medical parameters were documented for every subject. Exclusion criteria were pregnancy, latex and polyvinyl chloride allergy, claustrophobia, hypotension, history of vein thrombosis, chronic obstructive pulmonary disease, epilepsy, cardiovascular and pulmonary diseases, and infectious diseases. Ten male and nine female volunteers were recruited, aged between 21 and 38 years with body-mass-indices from 17.2 to 32.5.

PPE suits Suit A: TychemR F overall whole-body (DuPont de Nemours and Company, 3M, Austria) suit including socks with a reusable light hood VersafloTM S-655 (3M, Austria) and an external 3M JupiterTM Powered Air Turbo Unit (3M Austria) providing head-only positive pressure.

Suit B: 3MTM JS-series Typ 3 Chemical and Respiratory Protective Suit (CRPS, 3M, Austria) with integrated respirator 3M Jupiter JP-ER-03 Powered Air Purifying Turbo (3M, Austria) fixed as a rucksack generating whole-suit positive pressure.

With both suits, Sempercare surgical gloves (Sempermed, powder-free 150; Semperit, Austria) as the first layer, Ansell Sol-Vex gloves 37-900 (Ansell, Medical GBU, VWR, Austria) as a second layer and white rubber boots were worn. Gloves and boots were sealed to the suit using adhesive tape. Tests I and II were performed in a mock-up glove box providing a third layer of latex gloves.

Tests Four tests were repeatedly performed as well as an additional questionnaire on comfort and general condition before the tests started and after every four-test-series. Test I comprised correct assembly and position of coloured and numbered 2 mL tubes and screwcaps in a storage device to test fine motor skills, concentration and error rate. Test II checked the same skills in a different approach by pipetting different volumes of coloured water into a 96-well microliter plate according to a given pattern. Test III "d2 Test of Attention" is a timed test of selective attention and a standardized refinement of a visual cancellation. In response to the discrimination of similar visual stimuli, the test measures processing speed, rule compliance, and quality of performance, allowing estimation of individual attention and concentration performance. Test IV investigated reaction time, mobility, speed and physical exercise by tapping touch sensors directed by signs on a screen (tapping test by talent-systems sportconsulting Gmbh, www.werthner.at). All subjects performed the tests after randomisation (www.randomizer.at) of the starting exercise. For example, subject one started with test I while subject two started with test II at the same time. After ten minutes testing time and a five minute break, subject one carried on with test II and subject two with test I. After a five minute break, subject one started with test III while subject two performed test IV over a 10 minute period. Again after five minutes break, subject one continued with test IV and subject two with test III. Subjects documented their individual comfort and general condition in a structured questionnaire before the tests started and after every series of tests. All four tests were repeated 6 times at 22°C (6 hours total working time) on the first test day and four times at 28°C (4 hours total working time) on the second test day. Limiting factors for working conditions were ranked after every series from 1 to 10 on the questionnaire whereby ranking 10 was a reason for terminating the study. Heart rate (HR) was measured with a wireless heart rate monitor placed below the sternum directly on the skin (Garmin Forerunner 305) before and after the test series (data used for statistical analysis) and additionally recorded during the test series. Body temperature and body weight were measured as well as weight of the respective PPE for calculating dehydration and evaluation of heat stress.

ELIGIBILITY:
Inclusion Criteria:

* healthy, good physical and mental resiliance

Exclusion Criteria:

* pregnancy, latex and PVC allergy, claustrophobia, hypotension, vein thrombosis, COPD, epilepsy, cardiovascular and pulmonary diseases, and infectious diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Physical measurements: Heart rate at 22°C and 28°C in each suit with 19 participants | up to 2 months
Measurement of concentration (d2 Test) at 22°C and 28°C in each suit with 19 participants. | up to 2 months
  This test will be analysed by descriptive analysis.
Measurement of error rates at 22°C and 28°C in each suit with 19 participants | up to 2 months
  For both temperatures repeated measurements and analysis of variances (rmANOVA) to assess effects of working time as a within subject factor and suit (A, B) as a between subject factor on the amount of processed tubes and the amount of wrongly screwed or arranged tubes are performed.
Measurement of individual perception and wellbeing during all test series by individual questionnaires at 22°C and 28°C in each suit with 19 participants. | up to 2 months
  Questionnaire data are recorded 7 times at 22°C and 5 times at 28°C and analysed with descriptive statistics.
Physical measurements: Fluid loss at 22°C and 28°C in each suit with 19 participants. | up to 2 months
Physical measurements: Body temperature at 22°C and 28°C in each suit with 19 participants. | up to 2 months
Measurement of reaction time at 22°C and 28°C in each suit with 19 participants. | upt o 2 months
  This test will be analysed by descriptive analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Zatloukal, Prof., Principal Investigator — kurt.zatloukal@medunigraz.at
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loibner M, Hagauer S, Schwantzer G, Berghold A, Zatloukal K. Limiting factors for wearing personal protective equipment (PPE) in a health care environment evaluated in a randomised study. PLoS One. 2019 Jan 22;14(1):e0210775. doi: 10.1371/journal.pone.0210775. eCollection 2019. PMID 30668567